CLINICAL TRIAL: NCT00755989
Title: A Phase 3, Single-centered, Randomized, Double-blind, Placebo-controlled, Efficacy and Safety Trial of Morphine Sulfate Gel 0.1% in Patients With Stage 2-3 Wounds
Brief Title: Use of Morphine Gel Topically in Patients With Stage 2-3 Wounds
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study {I is no longer with banner Health, please remove this study from Banner Health's list.
Sponsor: Banner Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: morphine gel
Record Dates: First submitted 2008-09-18; First posted 2008-09-19 (Estimated); Last update posted 2025-07-20 (Actual); Status verified 2025-02

CONDITIONS: Wounds
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm Title 1 (Other): None available - study is no longer active.
  Interventions: Other: None available

INTERVENTIONS:
Other: None available
  Other Names: STudy is no longer active

SUMMARY:
Morphine gel applied topically to wounds will reduce wound pain and decrease patients use of oral and intravenous pain medications, therefore reducing side effects.

DETAILED DESCRIPTION:
Patients will be randomized to receive either placebo (versa base gel) or morphine gel to wound. Patients receiving morphine gel will have a decrease in pain score and use less oral/intravenous pain medications.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated consent form & HIPAA
* >/= 18 yo
* Single stage 2-3 wound evaluated by our wound care team
* Alert and oriented (thinking ability clear and intact, physician approval)
* English language proficiency, likely to be able to participate in all scheduled evaluations

Exclusion Criteria:

* Allergy to morphine, codeine, or versa base
* pts taking medications for acute condition, other than for the wound pain (can be taking chronic pain meds if current dose stable for past 3 mo)
* Patients with neuropathies
* Patients with respiratory conditions
* Patients that are pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-04; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Safety and efficacy with the use of morphine gel applied topically for pain control | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mary Whitmer, MSN,FNP, APRN BC-PCM, Principal Investigator — Banner Health
Locations (1):
- Banner Good Samaritan Medical Center, Phoenix, Arizona, United States